CLINICAL TRIAL: NCT05418270
Title: Anorexia and Personality Traits in Elderly Individuals
Acronym: APETI
Status: Completed | Type: Observational
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Sponsor
Other Study IDs: APETI
Record Dates: First submitted 2022-06-09; First posted 2022-06-14 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Anorexia; Personality; Aging; Chronic Disease
Keywords: anorexia; personality; aging; Chronic Disease
MeSH Terms: conditions — Anorexia; Chronic Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to evaluate the relationship between age-related anorexia and personality traits in elderly individuals with comorbidities.

DETAILED DESCRIPTION:
There is no study in the literature investigating the relationship between personality traits and age-related anorexia. The aim of this study is to evaluate the relationship between age-related anorexia and personality traits in elderly individuals with comorbidities.

ELIGIBILITY:
Inclusion Criteria:

* Being 65 years or older,
* Volunteering to participate in the study,
* Being conscious and not having communication problems,
* Having a Charlson comorbidity index of 1 or higher and/or a diagnosis of hypertension,
* Being fed orally.

Exclusion Criteria:

* oropharyngeal dysphagia,
* Presence of neurological or muscular disease that prevents swallowing,
* Being fed by nasogastric tube, percutaneous endoscopic gastrostomy or intravenous nutrition,
* Using drugs that affect appetite (corticosteroid, cancer chemotherapy digoxin, opioids, serotonin reuptake inhibitors, topiramate),
* Using appetizers (megestrol acetate, dronabinol, mirtazapine, growth hormone analogue),
* Having an active cancer disease,
* Major neuro-psychiatric disease (Alzheimer's, dementia, major depression, mania, psychosis, etc.),
* Presence of acute infection,
* Not having sufficient communication skills (Mini Mental Test score below 24 points).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: 65 years of age and older with chronic illness
Sampling Method: Non-Probability Sample
Enrollment: 310 (Actual)
Dates: Start 2022-06-02 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
relationship between anorexia and personality traits | 1 week
  relationship between anorexia and personality traits measured by Simplified Nutritional Appetite Questionnaire (SNAQ) and Five Factor Personality Inventory - Short Form scores

CONTACTS AND LOCATIONS:
Overall Officials: Elif Yıldırım Ayaz, M.D., Principal Investigator — Sultan Abdülhamid Training And Research Hospital
Locations (1):
- Sultan Abdülhamid Training and Research Hospital, Üsküdar, Istanbul, Turkey (Türkiye)